CLINICAL TRIAL: NCT06150131
Title: Combination of Supervised and Non-supervised Exercise After Lung Cancer Surgery
Brief Title: Exercise Intervention After Lung Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 281273
Record Dates: First submitted 2023-09-26; First posted 2023-11-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-09

CONDITIONS: Rehabilitation After Lung Cancer Surgery
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Supervised exercise one session per week, un-supervised exercise two sessions per week, for tree months, followed by three months without organized exercise.
  Interventions: Other: Exercise
- Control group (Other): Three months without organized exercise, followed by the same exercise as the Treatment group for three months.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Aerobic and strength exercise.
  Arms: Treatment group
Other: Exercise — Aerobic and strength exercise.
  Arms: Control group

SUMMARY:
A combination of supervised and un-supervised exercise in patients after lung cancer surgery is evaluated with regards to aerobic capacity, strength, physical activity and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Elective lung cancer surgery
* Ability to perform tests
* Able to communicate in Swedish
* Willing to participate in supervised exercise

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | 30 minutes
  Measuring the distance walked in 6 minutes.

SECONDARY OUTCOMES:
EORTC QLQ-C30/LC13 | 10 minutes
  Scale 0-100, for function scales higher is better, for symptom scales higher means more symptoms.
30 s chair stands test | 5 minutes
  Measuring the number of stands from a chair during 30 seconds.
OMPAQ | 2 minutes
  Categorical question on physical activity performed during the last month.
Actigraph GT3X | 7 days
  Accelerometer providing information about steps and time in different intensities of physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No